CLINICAL TRIAL: NCT03331809
Title: Influence of Two-handed Jaw Thrust on Postoperative Sore Throat in Patients Undergoing Double-lumen Endobronchial Tube Insertion
Brief Title: Two Handed Jaw-thrust on Postoperative Sore Throat After Double-lumen Endotracheal Tube Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-11-002
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-06

CONDITIONS: Lung Surgery
Keywords: intubation; pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Procedure: Conventional intubation
- Two-hand (Experimental)
  Interventions: Procedure: Two-handed jaw thrust

INTERVENTIONS:
Procedure: Two-handed jaw thrust — The assistant applied two-handed jaw thrust when intubating with double-lumen tube endotracheal tube.
  Arms: Two-hand
Procedure: Conventional intubation — The attending anesthesiologist provided intubation with double-lumen tube endotracheal tube without two-handed jaw thrust.
  Arms: Control

SUMMARY:
This investigation is planned to compare the incidence and severity of postoperative sore throat according to the use of two-handed jaw thrust maneuver in patients undergoing double-lumen endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients scheduled for double-lumen endotracheal intubation

Exclusion Criteria:

* Difficult airway
* Mallampatti scores greater than 3
* Recent sore throat
* Cervical spine disease
* History of head and neck surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative sore throat for postoperative 24 h | At 24 hr

SECONDARY OUTCOMES:
Number of participants with postoperative sore throat | At 1, 6, and 24 hr
Postoperative sore throat scores | At 1, 6, and 24 hr
  Visual anlogue scales will be used (10: most imaginable pain, 0: no pain).
Number of participants with postoperative hoarseness | At 1, 6, and 24 hr
Number of participants with postoperative shivering | At 1, 6, and 24 hr
Wound pain scores | At 1, 6, and 24 hr
  Visual anlogue scales will be used (10: most imaginable pain, 0: no pain).
Jaw discomfort scores | At 1, 6, and 24 hr
  Visual anlogue scales will be used (10: most imaginable pain, 0: no pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Keimyung University, Daegu, Non-US/Canada, South Korea

REFERENCES:
- [Derived] Park JJ, Huh H, Yoon SZ, Lim HJ, Go DY, Cho JE, Lee J, Park J, Kim HC. Two-handed jaw thrust decreases postoperative sore throat in patients undergoing double-lumen endobronchial intubation: A randomised study. Eur J Anaesthesiol. 2020 Feb;37(2):105-112. doi: 10.1097/EJA.0000000000001149. PMID 31860598